CLINICAL TRIAL: NCT00056238
Title: A Phase II Pilot Study of the Safety, Tolerability and Pharmacokinetics of Cerebril™ in Patients With Lobar Hemorrhage Related to Cerebral Amyloid Angiopathy
Brief Title: Cerebril™ in Patients With Lobar Hemorrhage Related to Cerebral Amyloid Angiopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-758003
Record Dates: First submitted 2003-03-07; First posted 2003-03-10 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: Stroke; Neurologic Diseases, General
Keywords: Neurologic Diseases (General); Hemorrhagic Stroke; Cerebral Amyloid Angiopathy; Cerebrovascular Accident
MeSH Terms: conditions — Stroke; Nervous System Diseases; Hemorrhagic Stroke; Cerebral Amyloid Angiopathy | interventions — NC 758; Pharmaceutical Preparations

INTERVENTIONS:
Drug: NC-758 (Anti amyloidotic [Aß] agent)

SUMMARY:
The main objective of this study is to evaluate the safety, tolerability and pharmacokinetics of Cerebril™ in Cerebral Amyloid Angiopathy (CAA) patients who have had lobar cerebral hemorrhage.

DETAILED DESCRIPTION:
Hemorrhagic Stroke due to CAA represents approximately 7% of all strokes.

The current phase II clinical study investigates the safety, tolerability, pharmacokinetic and pharmacodynamic profiles of the drug candidate in patients who have suffered lobar hemorrhages. The initial phase of the study is also aimed at determining the optimal dosing regimens for subsequent drug candidate efficacy trials. The trial is also evaluating the appearance of new cerebral hemorrhages on gradient-echo MRI scans, the amyloid ß (Aß) protein levels in the plasma and cerebrospinal fluid and the neurological and cognitive functions.

ELIGIBILITY:
Inclusion Criteria

* Patients must be 55 years of age or older.
* Males and females. Females must be of non-childbearing potential (i.e. surgically sterilized or at least one year post-menopausal).
* Diagnosis of possible or probable CAA based on the Boston Criteria for Diagnosis of CAA-Related Hemorrhage.
* Nonfatal lobar hemorrhage (defined as hemorrhage in the cerebral cortex and underlying white matter sparing the basal ganglia and thalamus) within previous five years diagnosed by CT or MRI scan.
* Patient has no intent to donate blood for 4 weeks after completion of the study.
* Signed informed consent.

Exclusion Criteria

* Other established causes of hemorrhage at the time of the index hemorrhage event. Exclusion causes include excessive anticoagulation (INR > 4.0), associated head trauma or ischemic stroke, CNS tumor, vascular malformation, vasculitis, and blood dyscrasia.
* Patient with a clinically significant and uncontrolled cardiovascular, renal, hepatic, pulmonary, gastrointestinal, endocrine, metabolic, ophthalmologic, hematological condition or other significant medical disease.
* Presence of any condition that could interfere with the interpretation of study results or compromise patient safety.
* Debilitated neurological state or other known disease likely to result in early death.
* Disability characterized by a modified Rankin score ≥ 4.
* ALT, ALP, AST or total bilirubin ≥ 1.5 the upper limit of normal ranges.
* Contraindications to MRI scan (e.g. cranial metallic implant, cardiac pacemaker, and severe claustrophobia).
* Allergy and/or hypersensitivity to analgesic agents used for the lumbar puncture (for patients undergoing lumbar puncture only).
* Allergy and/or hypersensitivity to any component of the study medication.
* Use of an investigational drug within 30 days prior to Screening visit.
* Use of warfarin or warfarin containing compounds and heparin or heparin containing compounds within 7 days prior to Baseline (Week 0) visit.
* Diagnosis of cystatin C amyloid angiopathy.
* Active alcohol and/or drug abuse.
* Inability to provide legal consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Greenberg, M.D., PhD., Principal Investigator — Massachusetts General Hospital; Co-sponsor: National Institute of Neurological Disorders and Stroke, Bethesda, MD, USA
Locations (5):
- United States (5):
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Gervais F, Chalifour R, Garceau D, Kong X, Laurin J, Mclaughlin R, Morissette C, Paquette J. Glycosaminoglycan mimetics: a therapeutic approach to cerebral amyloid angiopathy. Amyloid. 2001 Jul;8 Suppl 1:28-35. PMID 11676287
- [Background] M.C. Belanger, P. Krzywkowski, J. Paquette, M. Yu, C. Ramassamy, P. Tremblay, and F. Gervais. Development of Cerebral Amyloid Angiopathy in the TgCRND8 Mouse Model of Alzheimer's Disease. Data presented at the Society for Neuroscience, Orlando, FL, November 2002.